CLINICAL TRIAL: NCT03181178
Title: Effect of a Complementary Food Supplement on Growth and Morbidity of Ghanaian Infants (6 to 18 Months)
Brief Title: Effect of a Complementary Food Supplement on Growth and Morbidity of Ghanaian Infants
Acronym: TRIUMF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nevin Scrimshaw International Nutrition Foundation (Other)
Collaborators: University of Ghana (Other); University of Cape Coast (Other); Ajinomoto USA, INC. (Industry); Ghana Health Services (Other Government)
Responsible Party: Principal Investigator, Shibani Ghosh, Senior Scientist, Nevin Scrimshaw International Nutrition Foundation
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Ghana Trial
Record Dates: First submitted 2017-06-05; First posted 2017-06-08 (Actual); Last update posted 2018-03-01 (Actual); Status verified 2018-02

CONDITIONS: Growth Disorders; Infant Malnutrition; Micronutrient Deficiency; Protein Malnutrition; Morbidity;Infant
Keywords: Complementary food supplement; Protein quality and linear growth; Intervention targeting complementary foods and growth
MeSH Terms: conditions — Growth Disorders; Infant Nutrition Disorders; Kwashiorkor | interventions — Nutrition Assessment

STUDY DESIGN:
Intervention Model Description: The study has three intervention arms and one cross sectional growth monitoring follow up group.
Who Masked: Participant
Masking Description: Single blind cluster randomized trial - all participants in a community received the same treatment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- KokoPlus and Nutrition Education (Active Comparator): Macro-micronutrient complementary food supplement and Nutrition Education
  Interventions: Dietary Supplement: Macro-micronutrient complementary food supplement; Behavioral: Nutrition education
- Micronutrient and Nutrition Education (Active Comparator): A micronutrient powder and Nutrition Education
  Interventions: Dietary Supplement: A micronutrient powder; Behavioral: Nutrition education
- Nutrition Education Only (Active Comparator): Nutrition Education
  Interventions: Behavioral: Nutrition education
- Growth Monitoring Only (No Intervention): Growth monitoring

INTERVENTIONS:
Dietary Supplement: Macro-micronutrient complementary food supplement — This intervention provided a 15 g complementary food supplement called KokoPlus with nutrition education
  Arms: KokoPlus and Nutrition Education
Dietary Supplement: A micronutrient powder — This intervention provided a 1 g micronutrient powder with nutrition education
  Arms: Micronutrient and Nutrition Education
Behavioral: Nutrition education — This intervention provided nutrition education sessions
  Arms: KokoPlus and Nutrition Education; Micronutrient and Nutrition Education; Nutrition Education Only

SUMMARY:
Prevention of malnutrition in infants and children requires access and intake of nutritious food starting at birth with exclusive breastfeeding for the first 6 months of life, breastfeeding in combination with complementary foods from 6-24 months of age, access to clean drinking water and sanitation, access to preventive and curative health care (including prenatal).

In Ghana, the Demographic and Health Survey of 2014 reports rates of stunting, wasting and underweight in children aged 0-59 months are 28%, 14% and 9% respectively. Furthermore, height for age starts dropping from age 4-6 months with children aged 6-23 months being more likely to be stunted (40%) than those below 6 months (4%). Infant and young child feeding data show that for breast-fed children ranging from 6 months through 35 months of age, cereals are predominantly the first foods introduced in the diet (6-8 months of age). As the child grows older, consumption of fruits rich in Vitamin A, other fruits and vegetables and meat, fish, poultry and eggs are reported by the mothers. The Demographic and Health Survey (DHS) found that the proportion of breast fed children aged 6-23 months who received a recommended variety of foods the minimum number of times per day increases with child's age from 28% in children 6-8 months to 50% in children aged 18-23 months.

The study objective is to examine the effect of providing a macro- and micro-nutrient fortified complementary food supplement (KokoPlusTM) on growth and nutritional status of Ghanaian infants.

DETAILED DESCRIPTION:
The current study is a cluster randomized single blind intervention design study with three study arms that aimed to examine the effect of providing a macro- and micro-nutrient fortified complementary food supplement (KokoPlus) for a period of 12 months (starting at 6 months of age) on growth and nutritional status of Ghanaian infants at 18 months of age. KokoPlus was formulated using linear programming methodology based on formative and market analysis research findings.

The subjects in this cluster-randomized trial are from communities in three districts of the Central region in Ghana with high rates of moderate and severe acute malnutrition. A total of 38 communities will be randomly assigned to one of three groups using block randomization and another 11 (randomly selected) will be followed cross sectionally as part of a fourth/non intervention group (growth monitoring).

The total sample size is 1204. Sample size calculations were based on two outcome measures: expected reduction in diarrheal morbidity and growth (improvements in height-for-age). Sample size estimates for detecting a 0.5 cm change in height in children provided a caloric and non caloric micronutrient supplement using a design effect of 2, power of 0.80, alpha of 0.05 and assuming an attrition rate of 15%, the required sample size per group was 301.

Mother-infant pairs will be recruited between infant age of 0 to 3 months to participate in monthly nutrition educations sessions and to encourage the women to continue exclusive breast feeding across all three groups. At 6 months of age, infants in each of the three groups were enrolled into the intervention study (upon receipt of informed consent). Data collection involves baseline, midline and endline measurements in the infants at 6, 12 and 18 months of age. In addition, participating mother-infant pairs will be visited weekly for delivery of the supplements and for morbidity monitoring and monthly for the measurement of anthropometry. Anthropometric measurements include: length (Infant/Child Shorr Height Board; Weigh and Measure, LLC ), weight (Seca 874 digital scale ), mid-upper arm circumference (MUAC) (Child MUAC Tape; Weigh and Measure, LLC), subscapular and triceps skinfolds (Holtain skinfold caliper ),head and chest circumference.

Data collection at baseline, midline and endline included one venous sample (3ml) from the infant, HemoCue (Model 301) measurement to assess severe anemia (7 <g/dl) with appropriate referrals as mentioned earlier. Ethylenediaminetetracetic acid (EDTA) Vacutainers (BD ; catalog number 368841) for whole blood and plasma analyses and Trace Element Serum Separator Tube Vacutainers (BD; catalog number 368380) for serum analyses will be used for the sample collection with butterfly needles (21 or 23 gauge). Samples will be immediately placed in a super cooler tube rack and transported back to the lab within five hours where they were processed immediately. Questionnaires will be administered to assess socio-economic status, infant and young child feeding practices, morbidity (past week), household food security along with a 24 hour diet recall. Data was uploaded daily through cellular network, stored on Formhub and then Ona organization servers.

The primary outcome of the study is the change in length for age Z-score from 6 to 18 months of age in infants in the KokoPlus group versus Micronutrient powder group and the Nutrition Education group. Data calculations included estimating anthropometric indices using the WHO (World Health Organization) 2006 growth reference charts using the WHO macro in STATA (18), computing the USAID Food and Nutrition Technical Assistance (FANTA) household insecurity access scores (HFIAS) (19) maternal body mass index (BMI), dietary diversity scores (20), and re-coding variables as required to binary and accounting for missing. Infant anthropometric indices calculated include length for age (LAZ) Z- score, weight for age Z-score (WAZ) and weight for length (WLZ score).

All analyses are intent to treat. Descriptive statistics (means, medians, standard deviations and standard errors) were computed. To verify the randomization assumption, any differences in mean values at baseline across three groups were tested using linear mixed effects regression analyses accounting for clustering. The effect of the supplement (KokoPlus, Micronutrients and Nutrition Education group) on different dependent variables across the intervention period will be tested using mixed effects regression analyses accounting for clustering and repeated measures. The dependent variables tested included change in LAZ between baseline and endline (primary outcome), change in LAZ on a monthly basis (primary outcome 2), change in WAZ, WLZ, serum hemoglobin (unadjusted and adjusted for inflammation), serum ferritin (unadjusted and adjusted for inflammation), serum zinc, serum cortisol, serum insulin growth factor-1 (IGF-1), serum retinol binding protein, C-reactive protein and alpha glycoprotein, prevalence of acute and chronic infection.

A cross-sectional assessment (anthropometry) will be conducted at baseline, midline and endline in 301 infants that are randomly selected from another set of communities (to be identified based on the same community selection criteria). These infants will not be followed longitudinally and the only measurements to be collected include weights and heights. Informed consent procedures will be similar to the three intervention arms. This group is a reference group only and cannot be included in any comparative analysis.

Monitoring of groups that receive a supplement will happen weekly. Compliance will be defined based on the number of supplement packets that are consumed per week. To assure that the mothers are compliant in using the supplement, they will be asked to return the empty supplement packages at the end of the week. Optimal compliance will be defined as consumption of at least 50% of the weekly samples. Supplements will be provided in plastic or paper bags with a clearly labelled household ID (identity number). Compliance and dose response to compliance will be reviewed in existing studies to determine minimum compliance required.

ELIGIBILITY:
Inclusion Criteria:

1. Non pre-term
2. Singleton birth
3. Exclusively or predominantly breast fed up to time of recruitment
4. Parents planning to live in community for a period of 12 months and willing to participate in the trial for the entire period
5. Receive informed consent from both parents and/or caregivers or from mother alone if single

Exclusion Criteria:

1. Severely anemic (<7 g/dl) (to be referred to Community Health Post (CHP) for routine care on anemia as recommended by Ghana Health Service)
2. Severely malnourished (MUAC <110 mm) (to be referred to CHP with Community-based Management of Acute Malnutrition (CMAM) protocol) and/or use of CMAM protocol or below -2 standard deviations (SD) weight for age Z score

Ages: 6 Months to 6 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1204 (Actual)
Dates: Start 2013-02 (Actual); Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Change in monthly length for age Z-score (monthly LAZ) | Measured on a monthly basis until 18 months of age
  Change in length for age Z-score from 6 months to 18 months of age.

SECONDARY OUTCOMES:
Change in Serum Hemoglobin | Baseline (6 months), Midline (12 months of age), Endline (18 months of age)
  Change in serum hemoglobin from baseline to endline (6 months to 18 months)
Change in Serum retinol binding protein | Baseline (6 months), Midline (12 months of age), Endline (18 months of age)
  Change in serum retinol binding protein from baseline to endline (6 months to 18 months)
Change in serum transferrin receptors | Baseline (6 months), Midline (12 months of age), Endline (18 months of age)
  Change from baseline to endline (6 months to 18 months)
Change in serum ferritin | Baseline (6 months), Midline (12 months of age), Endline (18 months of age)
  Change from baseline to endline (6 months to 18 months)
Change in serum zinc | Baseline (6 months), Midline (12 months of age), Endline (18 months of age)
  Change from baseline to endline (6 months to 18 months)
Change in Weight for age Z-score | Measured at baseline and then on a monthly basis for the duration of the intervention (12 months)
  This is the change in weight for age Z-score from 6 months to 18 months of age
Change in Weight for height Z-score | Measured at baseline and then on a monthly basis for the duration of the intervention (12 months)
  This is the change in weight for length Z-score from 6 months to 18 months of age
Prevalence of diarrhea | Measured at baseline and then in a weekly surveillance for the duration of the intervention (12 months or 52 weeks)
  Prevalence of diarrhea over a 12 month period (duration of intervention)
Prevalence of upper respiratory infections | Measured at baseline and then in a weekly surveillance for the duration of the intervention (12 months or 52 weeks)
  Prevalence of respiratory infections over a 12 month period (duration of the intervention)
Change in serum C-reactive protein | Baseline (6 months), Midline (12 months of age), Endline (18 months of age)
  Change from baseline to endline (6 months to 18 months)
Change in serum alpha glycoprotein | Baseline (6 months), Midline (12 months of age), Endline (18 months of age)
  Change from baseline to endline (6 months to 18 months)
Change in Head Circumference for age | Measured at baseline and then on a monthly basis for the duration of the intervention (12 months)
  This is the change in head circumference for age from 6 months to 18 months of
Change in MUAC (Mid Upper Arm Circumference) | Measured at baseline and then on a monthly basis for the duration of the intervention (12 months)
  This is the change in MUAC for age from 6 months to 18 months of age
Change in Plasma Amino Acid levels | Baseline (6 months), Midline (12 months of age), Endline (18 months of age)
  This is the change in individual plasma amino acids from 6 months to 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Shibani Ghosh, PhD, Principal Investigator — Nevin Scrimshaw International Nutrition Foundation; Gloria Otoo, PhD, Principal Investigator — University of Ghana; Kwaku Tano-Debrah, PhD, Principal Investigator — University of Ghana

IPD SHARING:
Plan to Share IPD: No
There is no plan to share individual participant data to other researchers

REFERENCES:
- [Background] de Pee S, Bloem MW. Current and potential role of specially formulated foods and food supplements for preventing malnutrition among 6- to 23-month-old children and for treating moderate malnutrition among 6- to 59-month-old children. Food Nutr Bull. 2009 Sep;30(3 Suppl):S434-63. doi: 10.1177/15648265090303S305. PMID 19998866
- [Background] Pan American Health Organization. Guiding Principles for Complementary Feeding of the Breast Fed Child p37, 2003
- [Background] Ghana Statistical Service, Ghana Health Service, ICF Macro Ghana Demographic and Health Survey 2008, Accra, Ghana, p 512, 2009
- [Derived] Furuta C, Sato W, Murakami H, Suri DJ, Otoo GE, Tano-Debrah K, Ghosh SA. Changes of Plasma Amino Acid Profiles in Infants With a Nutrient-Fortified Complementary Food Supplement: Evidence From a 12-Month Single-Blind Cluster-Randomized Controlled Trial. Front Nutr. 2021 Sep 30;8:606002. doi: 10.3389/fnut.2021.606002. eCollection 2021. PMID 34660654